CLINICAL TRIAL: NCT02177461
Title: A PROBE (Prospective, Randomised, Open-Label, Blinded Endpoint) Trial to Investigate the Efficacy and Safety of Telmisartan 40-80mg Once Daily Compared With 10-20 mg Enalapril Once Daily Over a Period of 24 Weeks in Elderly Patients With Blood Hypertension
Brief Title: Telmisartan Compared With Enalapril in Elderly Patients With Blood Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502.317
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Enalapril; Clonidine

ARMS (4):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Enalapril (Active Comparator)
  Interventions: Drug: Enalapril
- Telmisartan + clonidine TTS1 (Experimental)
  Interventions: Drug: Telmisartan; Drug: Clonidine
- Enalapril + clonidine TTS1 (Active Comparator)
  Interventions: Drug: Enalapril; Drug: Clonidine

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan; Telmisartan + clonidine TTS1
Drug: Enalapril
  Arms: Enalapril; Enalapril + clonidine TTS1
Drug: Clonidine
  Arms: Enalapril + clonidine TTS1; Telmisartan + clonidine TTS1

SUMMARY:
Study to assess the efficacy and tolerability of Telmisartan 40-80 mg once daily compared with enalapril 10-20 mg once daily in elderly patients with arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Sitting systolic blood pressure (SBP) ≥ 160 mmHg and any diastolic blood pressure (DBP) (safety maximum of sitting DBP 110 mmHg), measured by manual cuff sphygmomanometer at the end of the wash-out period
* Written informed consent

Exclusion Criteria:

* Secondary hypertension
* Malignant hypertension (retinal haemorrhage, exudates or papillary oedema)
* Clinically significant sodium depletion as defined by serum sodium level < 130 mEq/L, clinically significant hyperkaliemia as defined by serum potassium level > 5.5 mEq/L, clinically significant hypokaliemia as defined by serum potassium level < 3.0 mEq/L
* Atrial fibrillation or frequent ventricular ectopic beats or other arrhythmias which could interfere with the cardiac rhythm
* Heart rate < 50 bpm
* Congestive heart failure (CHF) (NYHA (New York Heart Association) functional class CHF III-IV)
* Angina pectoris or myocardial infarction
* Cardiac surgery within the past 3 months prior to start the wash-out period
* Stroke within the past 6 months prior to start the wash-out period
* Renal insufficiency defined as creatininaemia > 2mg/dl
* Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post renal transplant
* Liver insufficiency, defined as bilirubinaemia > 2mg/dl and AST (aspartate aminotransferase) or ALT (alanine-aminotransferase) > twice the upper normal range
* Clinically significant metabolic and endocrine disease
* Autoimmune disease
* Previous history of angioedema
* Body mass index > 30kg/m2
* Arm circumference > 32 cm
* Any condition that may be likely to compromise the trial (alcohol or drug abuse, disability illness, etc.)
* Concomitant therapy with antihypertensive drugs non-permitted by protocol, or present use of tricyclic antidepressant, corticosteroids or drugs known to affect blood pressure
* Investigational drug treatment within the past 30 days before the enrolment or concurrent participation to any other trial
* Sensitivity, significant adverse reaction or contraindications to the study drugs (telmisartan, enalapril, clonidine TTS)
* Predictable lack of patient co-operation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 374 (Actual)
Dates: Start 2000-04; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in 24-hours mean systolic blood pressure (SBP) (ABPM - ambulatory blood pressure measurement, 24 hours mean represents the average of 24 hourly mean values) | Baseline and week 8

SECONDARY OUTCOMES:
Comparison of SBP ABPM tracing profile | Week 8 and 24
Changes from baseline in trough cuff (sphygmomanometer) SBP | Baseline, week 8 and 24
Smoothness index in comparison with baseline | Baseline, week 8 and 24
Number of responders | Week 8 and 24
Number of controlled responders | Week 8 and 24
Incidence of adverse events | 24 weeks
Number of patients who withdraw due to adverse events | 24 weeks